CLINICAL TRIAL: NCT00657228
Title: Intravenous Heparin as an Adjunct for the Treatment of Anaphylactic/Anaphylactoid Reactions in the Emergency Department
Brief Title: Intravenous Heparin as an Adjunct for the Treatment of Anaphylactic Reactions in an Emergency Department
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study did not start.
Sponsor: University of Missouri, Kansas City (Other)
Collaborators: Truman Medical Center (Other); Saint Luke's Hospital (Unknown); Emergency Physicians Foundation of KC (Unknown); American College of Emergency Physicians (Other)
Responsible Party: Ryan Jacobsen, M.D., Truman Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 07-58
Record Dates: First submitted 2008-04-09; First posted 2008-04-14 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2017-01

CONDITIONS: Anaphylaxis
Keywords: Anaphylaxis; Anaphylactoid reactions
MeSH Terms: conditions — Anaphylaxis | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Placebo Comparator): Standard treatment (epinephrine, corticosteroids, diphenhydramine, and H2 blockers) plus an equal volume bolus of normal saline after the first doses are administered.
  Interventions: Drug: Saline
- 1 (Experimental): Standard therapy plus a one-time bolus of heparin at 80 U/kg (maximum dose of 10,000 Units) given immediately after the first doses of standard treatment.
  Interventions: Drug: Intravenous heparin

INTERVENTIONS:
Drug: Intravenous heparin — Intravenous heparin as an adjunct for the treatment of anaphylactic/anaphylactoid reactions in the Emergency Department.
  To determine if a single bolus of intravenous unfractionated heparin (in conjunction with standard therapy) given to patients with anaphylactic/anaphylactoid reactions results in a faster time to recovery when compared to standard therapy alone.
  Arms: 1
Drug: Saline — Standard treatment (epinephrine, corticosteroids, diphenhydramine, and H2 blockers) and saline.
  Arms: 2

SUMMARY:
To determine if intravenous unfractionated heparin (with standard therapy) for treatment of anaphylaxis results in faster time to recovery.

DETAILED DESCRIPTION:
Anaphylaxis is a potentially life-threatening entity that requires both immediate recognition and aggressive treatment. Although anaphylaxis is infrequent, comprising only 1% of approximately 1.03 million visits to the ED each year that are related to allergic reactions, it is none the less a generally under-recognized and under-treated disease, that is worthy of study due to the potential for a fatal outcome. Recently, there has been renewed interest in a commonly used and inexpensive drug (heparin) as a novel component of therapy for anaphylactic/anaphylactoid reactions. Heflin eft al. induced anaphylactoid reactions in pigs and compared intravenous unfractionated heparin in one treatment arm to standard therapy (intravenous epinephrine and diphenhydramine) versus placebo. The study revealed that heparin rapidly reversed the shock similar to that of standard emergency treatment. Of course this single study done in pigs will not change practice, but it does warrant further investigation into the role that heparin plays in anaphylaxis in humans.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* English speaking
* Meets one of the above definitions of anaphylaxis
* Signs/symptoms onset <12 hours will get epinephrine or will not get epinephrine because of contraindication to epinephrine administration.

Exclusion Criteria:

* History of Intracranial Hemorrhage at anytime
* Known Cerebral Vascular Lesion (i.e. Aneurysm, Arteriovenous malformation)
* Ischemic CVA within the last 3 months
* Suspected Aortic Dissection
* Active Bleeding
* Known Bleeding/Clotting Disorder
* Closed Head Trauma within the past 3 months
* Major Surgery (Abdominal/Thoracic) within the last 3 weeks
* Active GI Bleeding
* Currently taking Warfarin
* Allergy to Heparins
* History of Heparin-induced Thrombocytopenia (AHA contraindications to fibrinolytic therapy 2005, Micromedix 2007)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-12; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Time to improve to a severity score of 1 or complete resolution of signs/symptoms. | 6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Jacobsen, MD, Principal Investigator — Truman Medical Center; Stefanie Ellison, MD, Principal Investigator — Truman Medical Center
Locations (2):
- United States (2):
  - Truman Medical Center ED, Kansas City, Missouri
  - St. Luke's Hospital ED, Kansas City, Missouri

REFERENCES:
- [Background] Sampson HA, Munoz-Furlong A, Campbell RL, Adkinson NF Jr, Bock SA, Branum A, Brown SG, Camargo CA Jr, Cydulka R, Galli SJ, Gidudu J, Gruchalla RS, Harlor AD Jr, Hepner DL, Lewis LM, Lieberman PL, Metcalfe DD, O'Connor R, Muraro A, Rudman A, Schmitt C, Scherrer D, Simons FE, Thomas S, Wood JP, Decker WW. Second symposium on the definition and management of anaphylaxis: summary report--Second National Institute of Allergy and Infectious Disease/Food Allergy and Anaphylaxis Network symposium. J Allergy Clin Immunol. 2006 Feb;117(2):391-7. doi: 10.1016/j.jaci.2005.12.1303. PMID 16461139
- [Background] Greenberg MR. Response to: Heparin reverses anaphylactoid shock in a porcine model. Ann Emerg Med. 2007 Apr;49(4):541-2; author reply 542. doi: 10.1016/j.annemergmed.2006.09.033. No abstract available. PMID 17371711
- [Background] Heflin CR, Brewer KL, Hack JB, Meggs WJ. Heparin reverses anaphylactoid shock in a porcine model. Ann Emerg Med. 2006 Aug;48(2):190-3. doi: 10.1016/j.annemergmed.2006.03.029. Epub 2006 Jun 22. PMID 16857468
- [Background] Gaeta TJ, Clark S, Pelletier AJ, Camargo CA. National study of US emergency department visits for acute allergic reactions, 1993 to 2004. Ann Allergy Asthma Immunol. 2007 Apr;98(4):360-5. doi: 10.1016/S1081-1206(10)60883-6. PMID 17458433
- [Background] Brown SG, Mullins RJ, Gold MS. Anaphylaxis: diagnosis and management. Med J Aust. 2006 Sep 4;185(5):283-9. doi: 10.5694/j.1326-5377.2006.tb00619.x. PMID 16948628